CLINICAL TRIAL: NCT00500799
Title: Role of the Cortical Medial Frontal Areas in Blepharospasm
Brief Title: Brain Changes in Blepharospasm
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070191; 07-N-0191
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-14

CONDITIONS: Blepharospasm
Keywords: Transcranial Magnetic Stimulation (TMS); Blink Reflex; Blepharospasm; Healthy Volunteer; HV
MeSH Terms: conditions — Blepharospasm

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the role of certain areas of the brain in blepharospasm, a type of dystonia (abnormality of movement and muscle tone) that causes unwanted or uncontrollable blinking or closing of the eyelids. The study will compare brain activity in healthy volunteers and in people with blepharospasm to find differences in the brain that may lead to better treatments for dystonia.

Healthy volunteers and people with blepharospasm who are 18 years of age and older may be eligible for this study. All candidates are screened with a medical history. People with blepharospasm also have a physical examination and blepharospasm rating.

Participants undergo transcranial magnetic stimulation (TMS) and electromyography (EMG) in two 4-hour sessions, separated by 1 to 7 days.

TMS

A wire coil is held on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in muscles of the face, arm or leg. During the stimulation, subjects may be asked to tense certain muscles slightly or perform other simple actions. Repetitive TMS involves repeated magnetic pulses delivered in short bursts of impulses. Subjects receive 60 pulses per minute over 15 minutes.

EMG

Surface EMG is done during TMS to measure the electrical activity of muscles. For this test, electrodes (small metal disks) are filled with a conductive gel and taped to the skin of the face....

DETAILED DESCRIPTION:
Objectives

This proposal will evaluate the role of an increase in excitability of the orbicularis oculi (OO) muscle representation in the medial frontal areas (supplementary motor areas, SMA) and anterior rostral cingulate: M3) in excessive blinking in patients with benign essential blepharospasm (BEB). We hypothesize that:

1. at rest, the decrease of the MEP after 15 minutes of 1Hz rTMS, targeting the SMA-M3, is more prominent in patients with BEP than in healthy control subjects,
2. at rest, the decrease of the MEP after 15 minutes of 1Hz rTMS targeting M1, is almost the same in patients with BEP and in healthy control subjects,
3. at rest, sICI of OO muscle will be decreased and ICF increased after stimulation of the SMA-M3 facial cortical area, in patients with BEP compared to healthy control subjects,
4. at rest sICI and ICF of the OO muscle will be the same after stimulation of the M1 facial area in patients with BEP and healthy control subjects,
5. in healthy control subjects facilitation of the MEPs evoked from M1 is more prominent during voluntary blinking,
6. in healthy control subjects facilitation of the MEP evoked from SMA-M3 is more prominent during involuntary blinking,
7. in patients with BEB there is facilitation of MEPs evoked from M1 and SMA-M3 during voluntary and involuntary blinking.
8. it is possible to evoke consistent and reproducible motor evoked responses (MEP) in the orbicularis oculi (OO) muscles by stimulating the two main cortical representations of upper facial region: in the medial frontal wall (SMA and cingulate cortex - its rostral part, M3) and in the primary motor cortex (M1) with transcranial magnetic stimulation (TMS).

Study population

36 patients with BEB but without severe forceful closure of eyelids, 36 normal volunteers.

Study design

Subjects will have 3 visits:

Visit 1: screening and blepharospasm score

Visit 2: stimulation of the OO muscle representation in SMA-M3 using low frequency rTMS (1Hz) with the Hesed coil (designed to stimulate deep brain).

Visit 3: stimulation of the OO muscle representation in M1 using low frequency rTMS (1Hz) using a standard eight-shaped coil.

Visits 2 and 3: single pulse TMS will be used to evoke MEPs from OO muscles. Paired pulse TMS will be used to assess sICI from OO muscles. The order of visits 2 and 3 will be randomly assigned.

Outcome measures

The main outcome measures will be the sizes of OO muscle MEPs and the amount of sICI assessed before and after 15 minutes of low frequency rTMS. The secondary outcome measures will be the sizes of OO muscle MEPs assessed before and during voluntary and involuntary blinks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers (aged 18 or older) who are willing to participate.
* Patients (aged 18 and older) with benign essential blepharospasm

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Subjects with a history of neurological or psychiatric disorder, current use or a history of alcohol or drug abuse, psychiatric disorders requiring hospitalization or prolonged treatment, head injury with loss of consciousness, or epilepsy.
* Subjects receiving drugs acting primarily on the central nervous system

EXCLUSION CRITERIA FOR PATIENTS:

* Subjects with a history of neurological disorders other than blepharospasm
* Subjects with a history of a psychiatric disorder, current use or a history of alcohol or drug abuse, psychiatric disorders requiring hospitalization or prolonged treatment, head injury with loss of consciousness, or epilepsy.
* Subjects receiving drugs acting primarily on the central nervous system
* Subjects who have been treated with botulinum toxin injections within 3 months prior to their participation in the study
* Subjects who are taking any medication for dystonia at the time of the study
* Subjects with severe forceful closure of eyelids, subjects scoring more than 20 on the Blepharospasm Disability scale (Lindeboom et al., 1995).
* Patients for whom participation in the study would, in the opinion of the investigators, cause undue stress or excessive apprehensiveness will also be excluded. The reason for that is that, in some patients, any stressful situation (like a medical exam or experiment) may cause a strong increase in the involuntary blink rate leading to a severe functional discomfort.

The following exclusion criteria are due to the use of transcranial magnetic stimulation and repetitive transcranial magnetic stimulation up to 1Hz (Hallett 1999) for healthy volunteers and patients:

* Subjects with cardiac pacemakers, intracardiac lines, implanted medication pumps.
* Subjects with eye, blood vessel, cochlear, or eye implants.
* Subjects with increased intracranial pressure as evaluated by clinical means
* Subjects with metal in the cranium
* Subjects with dental braces (but dental fillings are not a problem), metal fragments from occupational exposure or surgical clips in or near the brain.
* Subjects with a personal or family history of hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2007-07-09; Study Completion 2009-04-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker RS, Andersen AH, Morecraft RJ, Smith CD. A functional magnetic resonance imaging study in patients with benign essential blepharospasm. J Neuroophthalmol. 2003 Mar;23(1):11-5. doi: 10.1097/00041327-200303000-00003. PMID 12616082
- [Background] Cunnington R, Iansek R, Thickbroom GW, Laing BA, Mastaglia FL, Bradshaw JL, Phillips JG. Effects of magnetic stimulation over supplementary motor area on movement in Parkinson's disease. Brain. 1996 Jun;119 ( Pt 3):815-22. doi: 10.1093/brain/119.3.815. PMID 8673493
- [Background] Gerschlager W, Siebner HR, Rothwell JC. Decreased corticospinal excitability after subthreshold 1 Hz rTMS over lateral premotor cortex. Neurology. 2001 Aug 14;57(3):449-55. doi: 10.1212/wnl.57.3.449. PMID 11502912